CLINICAL TRIAL: NCT06018987
Title: A Multicenter, Evaluator-blinded, Randomized, Delayed Treatment Control Group Study of the Safety and Effectiveness of HAC 20L for the Correction of Moderate to Severe Nasolabial Folds
Brief Title: A Study to Assess Adverse Events and Effectiveness of HAC 20L Injections in Adult Participants for the Treatment of Nasolabial Folds
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: M21-833
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Nasolabial Folds
Keywords: HAC 20L; AGN-8010; Nasolabial Folds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1: Treatment Group (Experimental): Participants will receive subdermal injection of HAC20L to the nasolabial folds on Day 1 followed by an optional touch-up treatment on Day 30 if applicable. Participants will then be eligible to receive optional repeat treatment at Month 12 if applicable.
  Interventions: Device: HAC 20L
- Cohort 1: Control Group (Other): Participants will not receive treatment for 6 months and then will be offered an optional delayed treatment of HAC 20L after completion of of Month 6 visit with an optional touch-up treatment offered 30 days after delayed treatment.
  Interventions: Other: No-Treatment Control
- Cohort 2: Treatment Group (Experimental): Participants will receive subdermal injection of HAC20L to the nasolabial folds on Day 1 followed by an optional touch-up treatment on Day 30 if applicable. Participants will then be eligible to receive optional repeat treatment at Month 12 if applicable.
  Interventions: Device: HAC 20L
- Cohort 2: Control Group (Other): Participants will not receive treatment for 6 months and then will be offered an optional delayed treatment of HAC 20L after completion of of Month 6 visit with an optional touch-up treatment offered 30 days after delayed treatment.
  Interventions: Other: No-Treatment Control

INTERVENTIONS:
Other: No-Treatment Control — Participants will not receive treatment for 6 months and then will be offered an optional delayed treatment of HAC 20L after completion of of Month 6 visit with an optional touch-up treatment offered 30 days after delayed treatment.
  Arms: Cohort 1: Control Group; Cohort 2: Control Group
Device: HAC 20L — Subdermal Injections
  Arms: Cohort 1: Treatment Group; Cohort 2: Treatment Group

SUMMARY:
Nasolabial folds (NLF) are the two skin folds that run from each side of the nose to the corners of the mouth. Prominent NLFs distort the contour of the midface, giving a fatigued and aged appearance. Soft tissue fillers can be used to reduce the depth of NLFs and restore a more youthful appearance. The purpose of this study is to evaluate how safe and effective HAC 20L is in the correction of moderate to severe NLF in adult participants.

HAC 20L is an investigational drug being developed for the treatment of NLF. There are 2 cohorts in this study. In each cohort participants are assigned to either the treatment group or no-treatment control group. There is a 1 in 3 chance that participants will be assigned to the no-treatment control group. Around 75 adult participants with moderate to severe NLF will be enrolled in the study at approximately 20 sites worldwide.

Participants in the treatment group will receive an injection of HAC 20L to the NLF on Day 1 in Cohort 1 and Cohort 2 with the option of re-treatment after completion of Month 12 visit. The control group will receive no treatment but will be offered an optional HAC 20L treatment after 6 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be examined by completing effectiveness questionnaires by the subjects, evaluating investigator (EI) and central reviewers as well as monitoring safety assessments such as vital signs, blood tests, injection site responses and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Has moderate or severe NLFs (NLFSS score 2 or 3) on each NLF based on EI's live assessment (both NLFs must qualify and need to have the same score).
* General good health, in the opinion of the TI, and no known current COVID 19 disease or previous COVID-19 disease-related symptoms within 30 days.

Exclusion Criteria:

* Atrophic skin in the facial area that makes it unsuitable for injection.
* History of anaphylaxis or history or presence of multiple severe allergies, including allergy to antiseptic solution, lidocaine (or any amide-based anesthetics), HA products, human recombinant collagen, bovine or porcine collagen products, gram positive bacterial proteins (including Streptococcal protein) or to any of the excipients.
* Prior fat injection or permanent implants (e.g., polymethylmethacrylate, silicone, polytetrafluoroethylene) anywhere in the face, or is planning to be implanted with any of these products at any time during the study.
* Received semipermanent soft-tissue filler treatment (e.g., calcium hydroxyapatite, poly-L-lactic acid) in the face below the orbital rim within 24 months before enrollment, or is planning to be implanted with any of these products at any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Responder Status Based on Evaluating Investigator's (EI's) Live Assessment of Nasolabial Folds (NLF) Severity using the Nasolabial Fold Severity Scale (NLFSS) | Month 6
  The NLFSS is a 5-point photonumeric scale used by the EI to assess the severity of each NFL where 0 = None and 4 = Extreme. A responder is defined as a participant who shows at least 1-point improvement on the NLFSS from baseline on both sides.
Number of Participants with Adverse Events (AEs) | Month 16
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this device

SECONDARY OUTCOMES:
Change from Baseline on the Overall Score of FACE-Q-Appraisal of Lines: Nasolabial Folds Questionnaire | Baseline to Month 6
  The FACE Q-Appraisal of lines: Nasolabial Folds consists of 5 questions to assess how much the participants has been bothered by various aspects of NLFs in the past week where 1 = not at all and 4 = extremely.
Percentage of Participants Achieving Responder Status Based on Evaluating Investigator's Assessment of Global Aesthetic Improvement on the NLF Area using the Global Aesthetic Improvement Scale (GAIS) | Month 6
  The GAIS will assess global aesthetic improvement of the NLF area by comparing the frontal and side view photographs taken at baseline where -2 = Much Worse and 2 = Much Improved. A responder is defined as achieving "improved" or "much improved".
Percentage of Participants Achieving Responder Status Based on Participant's Assessment of Global Aesthetic Improvement in the NLF Area Using the GAIS | Month 6
  The GAIS will assess global aesthetic improvement of the NLF area by comparing the frontal and side view photographs taken at baseline where -2 = Much Worse and 2 = Much Improved. A responder is defined as achieving "improved" or "much improved".

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- Germany (10):
  - Hautok and Hautok-cosmetics /ID# 254549, Munich, Bavaria
  - Dermatologische Gemeinschaftspraxis Mahlow /ID# 232366, Blankenfelde-Mahlow, Brandenburg
  - MediCorium Zentrum fuer Dermatologie und Aesthetik /ID# 231403, Oberursel, Hesse
  - Hautzentrum Koeln /ID# 231406, Cologne, North Rhine-Westphalia
  - Privatpraxis Dr. Hilton & Partner /ID# 231401, Düsseldorf, North Rhine-Westphalia
  - CRS Clinical Research Services Berlin GmbH /ID# 240390, Berlin
  - Dermatologie am Luegplatz /ID# 233788, Düsseldorf
  - Universitaet Hamburg /ID# 231641, Hamburg
  - Noahklinik GmbH /ID# 231917, Kassel
  - Privatpraxis fuer Dermatologie und Aesthetik /ID# 231402, München

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M21-833